CLINICAL TRIAL: NCT01990794
Title: A 90-Day Cobalt Supplementation Study to Investigate the Cobalt Body Burden in Ten Healthy Adult Volunteers
Brief Title: 90-Day Cobalt Supplementation Study to Investigate the Cobalt Body Burden in Ten Healthy Adult Volunteers
Status: Completed | Type: Observational
Sponsor: Cardno ChemRisk (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103
Record Dates: First submitted 2013-11-12; First posted 2013-11-21 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Cobalt Biokinetics; Safety of Cobalt Dietary Supplementation
Keywords: Cobalt; Dietary Supplements; Hematological; Thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study Volunteers: Volunteers (males and females) were instructed to take the cobalt dietary supplement in the morning according to the manufacturer's label, which suggested a serving of 1 mg cobalt (~2 mL) daily "in water or juice as maintenance." Dietary supplementation lasted for approximately three months.

SUMMARY:
The purpose of this study is to investigate steady-state cobalt levels following dietary supplementation for 90 days with 1 mg cobalt/day (as cobalt chloride in solution) in healthy adult volunteers.

DETAILED DESCRIPTION:
Over the counter cobalt (Co) dietary supplements are available for sale in the United States, but little is known regarding their clinical effects and biokinetic distribution and body burden with long-term use. This study assessed blood kinetics, steady-state levels, biochemical responses, and clinical effects in five adult males and five adult females who voluntarily ingested approximately 1.0 mg Co/day of a commercially available Co supplement over a three month period. Volunteers were instructed to take the Co-dietary supplement in the morning according to the manufacturer's label. Blood samples were collected and analyzed for a number of biochemical parameters before, during, and after dosing. Hearing, vision, cardiac, and neurological functions were also assessed in volunteers before, during, and after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years old.
* Subject able to understand and willing to sign a written informed consent form for the study.

Exclusion Criteria:

* Subject is unwilling to discontinue current multivitamins or other types of dietary supplements while on study
* Subject has a documented history of an allergy to cobalt
* Subject has a documented history of severe cardiac problems (e.g., congestive heart failure, myocardial ischemia within past 12 months, cardiomyopathy)
* Subject has a documented history of thyroid, kidney, or liver disease
* Subject has insulin-dependent diabetes
* Subject has a concurrent illness or personal stressor which in the opinion of the investigator may interfere with the subject's ability to perform the study's requirements.
* Subject has a total joint replacement (e.g., knee, hip, shoulder)
* Subject is pregnant or breastfeeding
* Subject is unwilling to follow protocol requirements
* Subject weight is less than 45 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers from work site and off work site
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Galbraith, MD, Principal Investigator — Cardno ChemRisk; David Galbraith, MD, Study Director — Cardno ChemRisk

REFERENCES:
- [Derived] Tvermoes BE, Unice KM, Paustenbach DJ, Finley BL, Otani JM, Galbraith DA. Effects and blood concentrations of cobalt after ingestion of 1 mg/d by human volunteers for 90 d. Am J Clin Nutr. 2014 Mar;99(3):632-46. doi: 10.3945/ajcn.113.071449. Epub 2014 Feb 5. PMID 24500148

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Volunteers
Started | 13
One Month Into Study | 10
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Our pair-wise comparisons had a power of 80% to detect a mean increase in RBC count of 0.34 million (sgma =0.2 million; n=5) and a mean increase of Hgb of 0.85 g/dL (sigma =0.5 g/dL; n=5), which are less than the minimum increases detected in the males that experienced polycythemia in Davis and Fields (1958).
Arm/Group | Study Volunteers
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years]
  Female Age (n=8) | 34 (10)
  Male Age (n=5) | 33 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Weight [Mean (Standard Deviation); unit: pounds (lbs)]
  Female weight (n=5) | 151 (20)
  Male weight (n=5) | 219 (53)

OUTCOME MEASURES:

1. Secondary Outcome: Albumin Bound Cobalt Fraction in Serum
Description: The fraction of albumin bound cobalt in serum was determined one to two weeks pre-dosing and on the day of the first dose before taking the supplement. Samples were also analyzed during the dosing period as follows: Day 4/5, Day 8/9, Day 14/16, Day 22/23, Day 29/30, Day 43/44, Day 57/58, Day 71/72, Day 88/90 and the fraction of albumin bound cobalt in serum was also determined at one and two weeks post-dosing.
Time Frame: Study volunteers will be followed for the duration of the study, an average of about 8 months for most volunteers
Population: Analysis was carried out on the first 12 participants of the study
Measure: Mean (Standard Deviation); unit: percentage of total blood cobalt
Groups:
- Albumin-Co Fraction: Summary of albumin-Co fraction (SEC large molecular Co fraction) in 12 volunteers participating in the cobalt supplementation study. The average for each volunteer is based on 2 to 11 blood draws during dosing.
Arm/Group | Albumin-Co Fraction
Number analyzed (Participants) | 12
percentage of total blood cobalt
  Subject 1 | 94.5 (4.9)
  Subject 2 | 95.2 (3.4)
  Subject 3 | 96.5 (2.9)
  Subject 4 | 93.2 (2.9)
  Subject 5 | 96.7 (2.7)
  Subject 6 | 95.6 (4.1)
  Subject 7 | 95.8 (2.5)
  Subject 8 | 95.7 (2.3)
  Subject 9 | 98.2 (2.7)
  Subject 10 | 94.9 (3.2)
  Subject 11 | 95.9 (2.9)
  Subject 12 | 96.7 (1.0)

2. Secondary Outcome: Effects on the Immune System
Description: Sensitivity to metals before and after cobalt supplementation was assessed by an in vitro lymphocyte transformation test (LTT) performed at week 0 and after three months of cobalt supplementation. The average proliferation rate for each metal treatment was normalized to individual proliferation rates of untreated control cells which generated a stimulation index (SI). According to the manufacture, the SI ranges from 0-15, with an SI from 2 to 4 indicated mild reactivity, from 5 to 8 indicated moderate reactivity, and >8 indicated high reactivity to the metal. The data is presented as the averaged normalized lymphocyte transformation response to each metal in men and women combined (n = 10).
Time Frame: 0 weeks and three months
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: units on a scale: stimulation index (SI)
Groups:
- SI Before Cobalt Supplementation; SI After Cobalt Supplementation: Volunteers (males and females) were instructed to take the cobalt dietary supplement in the morning according to the manufacturer's label, which suggested a serving of 1 mg cobalt (~2 mL) daily "in water or juice as maintenance." Dietary supplementation lasted for approximately three months. Metal sensitivity to metals was assessed before and after cobalt dosing by using an in vitro lymphocyte transformation test (LTT).
Arm/Group | SI Before Cobalt Supplementation | SI After Cobalt Supplementation
Number analyzed (Participants) | 10 | 10
units on a scale: stimulation index (SI)
  Normalized lymphocyte transformation response: Al | 1.79 (1.77) | 2.34 (3.0)
  Normalized lymphocyte transformation response: Co | 1.05 (0.32) | 1.44 (0.72)
  Normalized lymphocyte transformation response: Cr | 1.01 (0.38) | 1.43 (0.46)
  Normalized lymphocyte transformation response: Mo | 1.23 (1.21) | 2.31 (1.17)
  Normalized lymphocyte transformation response: Ni | 4.21 (3.62) | 4.32 (3.0)
  Normalized lymphocyte transformation response: V | 1.63 (0.82) | 1.86 (0.79)
  Normalized lymphocyte transformation response: Zr | 1.43 (0.56) | 1.41 (0.87)
  Normalized lymphocyte transformation response: Fe | 1.47 (0.91) | 1.82 (1.62)

3. Secondary Outcome: Hemoglobin Levels After 1, 2 and 3 Months of Dosing
Description: Blood chemistries assessed during the study included a lipid panel, comprehensive metabolic panel, creatine kinase-myocardial band, thyroid stimulating hormone, free thyroxine, and complete blood count with differential, total iron, and ferritin. Blood chemistries were assessed at one or two week pre-dose, pre-dose/ Day 1 before taking the supplement, Day 29/30, Day 57/58, Day 88/90 and one and two weeks post-dose.
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: Participants that completed three months of cobalt supplementation. Individual baseline values for the 1-wk predose draw and the day 1 (predose) draw were averaged together to give one baseline value.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Female Hgb: Hgb levels before, during and after dosing
- Male Hgb: Hgb levels before, during, and after dosing
Arm/Group | Female Hgb | Male Hgb
Number analyzed (Participants) | 5 | 5
g/dL
  Baseline (n = 5, 5) | 13.5 (0.43) | 14.9 (0.93)
  Days 29 and 30 (n = 5, 5) | 13.3 (0.50) | 14.8 (0.82)
  Days 57 and 58 (n = 5, 5) | 13.2 (0.37) | 15.1 (0.74)
  Days 88 and 90 (n = 5, 5) | 13.1 (0.31) | 14.9 (0.76)
  1 wk postdose (n = 5, 5) | 13.4 (0.75) | 14.9 (0.78)
  2 wk postdose (n = 5, 5) | 13.1 (0.61) | 15.0 (0.4)

4. Secondary Outcome: Changes in Audiological Function
Description: Audiologic assessments including pure tone threshold determination at frequencies ranging from 250 to 16000 Hz were performed with volunteers serving as their own baseline controls for receptive changes during the study (i.e., week 0, ~day 45, ~day 90). Audiologic assessments including a pure-tone threshold determination at frequencies that ranged from 250 to 16000 Hz were performed with volunteers serving as their own baseline controls for receptive changes during the study. Decreases in hearing were considered clinically significant when one of the following 3 American Speech-Language-Hearing Association criteria were met: 1) a ≥20-dB decrease in the pure-tone threshold at one test frequency, 2) a ≥10-dB decrease at 2 adjacent test frequencies, or 3) the loss of 3 consecutive test frequencies where responses were previously obtained.
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Baseline - Left; Baseline - Right; Study Midpoint - Left; Study Midpoint - Right; Study Completion - Left; Study Completion - Right: Comparison of hearing function in volunteers before, during, and after cobalt supplementation
Arm/Group | Baseline - Left | Baseline - Right | Study Midpoint - Left | Study Midpoint - Right | Study Completion - Left | Study Completion - Right
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
dB
  250 Hz | 10.0 (4.7) | 8.0 (6.3) | 9.0 (3.9) | 8.0 (6.7) | 7.5 (3.5) | 6.0 (5.7)
  500 Hz | 10.0 (4.1) | 6.0 (6.1) | 8.5 (4.7) | 7.5 (6.8) | 6.5 (4.7) | 5.5 (5.0)
  1000 Hz | 9.0 (3.2) | 7.5 (2.6) | 6.5 (4.1) | 5.0 (4.1) | 6.5 (4.7) | 7.5 (4.2)
  2000 Hz | 9.0 (5.7) | 9.5 (4.4) | 8.5 (6.7) | 9.5 (6.0) | 7.0 (6.8) | 7.5 (6.3)
  3000 Hz | 7.0 (7.5) | 8.5 (4.7) | 7.5 (6.8) | 8.0 (4.2) | 8.0 (7.5) | 5.0 (3.3)
  4000 Hz | 10.5 (9.0) | 6.0 (5.7) | 9.5 (10.1) | 6.0 (5.2) | 8.5 (10.5) | 7.5 (5.4)
  6000 Hz | 10.0 (8.5) | 12.0 (8.9) | 11.0 (9.1) | 11.0 (9.9) | 9.0 (6.9) | 10.0 (9.7)
  8000 Hz | 5.5 (7.6) | 10.0 (7.8) | 8.5 (8.8) | 7.5 (7.2) | 9.0 (7.1) | 7.5 (5.4)
  12,000 Hz | 9.5 (13.0) | 7.5 (10.1) | 8.5 (11.8) | 9.0 (8.1) | 9.5 (12.4) | 8.0 (7.9)
  16,000 Hz | 24.0 (21.2) | 25.5 (24.9) | 21.0 (22.6) | 25.0 (24.7) | 22.0 (20.0) | 24.0 (22.2)

5. Secondary Outcome: Changes in Cardiac Function
Description: Two-dimensional and Doppler echocardiographic examinations were used to assess cardiac anatomy, structure, and function during the study with volunteers serving as their own baseline controls for changes during the study (i.e., week 0, ~day 45, ~day 90).
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Prestudy; Study Midpoint; Study Completion: Comparison of left and right ventricular function in volunteers before and after cobalt supplementation
Arm/Group | Prestudy | Study Midpoint | Study Completion
Number analyzed (Participants) | 10 | 10 | 10
cm
  LVID (ed) (cm) | 4.77 (0.52) | 4.75 (0.55) | 4.65 (0.44)
  LVID (es) (cm) | 3.15 (0.38) | 2.97 (0.49) | 2.95 (0.55)
  RVID (ed) (cm) | 2.08 (0.46) | 2.02 (0.38) | 2.16 (0.35)
  Ao Root (ed) (cm) | 2.99 (0.38) | 3.03 (0.45) | 3.01 (0.44)
  IVS (ed) (cm) | 1.07 (0.19) | 1.06 (0.22) | 1.05 (0.13)
  IVS (es) (cm) | 1.40 (0.24) | 1.46 (0.24) | 1.48 (0.24)
  LVPWs (ed) (cm) | 0.94 (0.12) | 0.95 (0.11) | 0.99 (0.13)
  LVPWs (es) (cm) | 1.49 (0.19) | 1.47 (0.18) | 1.52 (0.15)
  LA (es) (cm) | 3.15 (0.21) | 3.34 (0.34) | 3.13 (0.44)

6. Secondary Outcome: Changes in Visual Function
Description: Ophthalmology studies included an assessment of visual acuity, slit lamp evaluations, and visual field testing. Retinal nerve fiber layer (RNFL) thickness and optic nerve head (ONH) were assessed using optical coherence tomography (OCT). Volunteers served as their own baseline controls for changes during the study (i.e., week 0, ~day 45, ~day 90).
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- Prestudy - Right; Study Midpoint - Right; Study Completion - Right: Values of the right eye for select ONH variables
- Prestudy - Left; Study Midpoint - Left; Study Completion - Left: Values of the left eye for select ONH variables
Arm/Group | Prestudy - Right | Prestudy - Left | Study Midpoint - Right | Study Midpoint - Left | Study Completion - Right | Study Completion - Left
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
mm^2
  Rim area (mm^2) | 1.29 (0.23) | 1.35 (0.23) | 1.38 (0.23) | 1.39 (0.29) | 1.31 (0.19) | 1.36 (0.25)
  Disc Area (mm^2) | 1.65 (0.30) | 1.73 (0.31) | 1.71 (0.33) | 1.74 (0.42) | 1.59 (0.20) | 1.63 (0.27)

7. Secondary Outcome: Changes in Neurological Function (Peroneal Motor Amplitude)
Description: Values of the sural sensory and peroneal motor variables. Volunteers served as their own baseline controls for changes during the study (i.e., week 0, ~day 45, ~day 90, and ~4-6 post-weeks).
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: Peroneal Motor Amplitude (mV)
Groups:
- Prestudy; Study Midpoint; Study Completion: Values of the sural sensory and peroneal motor variables
Arm/Group | Prestudy | Study Midpoint | Study Completion
Number analyzed (Participants) | 10 | 10 | 10
Peroneal Motor Amplitude (mV) | 5.1 (2.3) | 5.5 (2.3) | 5.6 (3.0)

8. Primary Outcome: Cobalt Whole Blood Concentrations
Description: The cobalt concentration in whole blood and serum was determined one to two weeks pre-dosing and on the day of the first day of dosing before taking the supplement. Samples were also analyzed during the dosing period as follows: Day 4/5, Day 8/9, Day 14/16, Day 22/23, Day 29/30, Day 43/44, Day 57/58, Day 71/72, and Day 88/90. Cobalt concentration in whole blood and serum was also determined at one, two, six, ten and 16 weeks post-dosing.
Time Frame: Before, during and after cobalt supplementation
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: µg Co/L
Groups:
- Female; Male: Volunteers (males and females) were instructed to take the cobalt dietary supplement in the morning according to the manufacturer's label, which suggested a serving of 1 mg cobalt (~2 mL) daily "in water or juice as maintenance." Dietary supplementation lasted for approximately three months.
Arm/Group | Female | Male
Number analyzed (Participants) | 5 | 5
µg Co/L
  Day 4/5 | 14.6 (8.2) | 7.4 (3.6)
  Day 8/9 | 33.9 (24.0) | 8.5 (6.9)
  Day 14/16 | 29.9 (22.0) | 13.8 (6.4)
  Day 22/23 | 25.6 (17.8) | 18.7 (11.3)
  Day 29/30 | 37.1 (24.8) | 19.3 (7.9)
  Day 43/44 | 35.9 (27.1) | 18.5 (10.5)
  Day 57/58 | 40.7 (28.1) | 20.3 (11.1)
  Day 71/72 | 37.1 (33.7) | 22.1 (11.5)
  Day 88/90 | 53.3 (45.3) | 20.4 (8.5)
  1 wk post | 22.2 (19.3) | 12.0 (6.3)
  2 wk post | 15.9 (13.3) | 8.7 (4.1)
  6 wk post | 9.7 (7.9) | 5.6 (2.9)
  10 wk post | 5.9 (5.4) | 3.9 (2.5)
  16 wk post | 1.1 (0.7) | 0.7 (0.2)

9. Secondary Outcome: White Blood Cell (WBC) Levels After 1, 2 and 3 Months of Cobalt Dietary Supplementation
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: thousand cells/µL
Groups:
- Female WBC: WBC levels before, during and after dosing
- Male WBC: WBC levels before, during, and after dosing
Arm/Group | Female WBC | Male WBC
Number analyzed (Participants) | 5 | 5
thousand cells/µL
  Baseline (n = 5, 5) | 6.46 (0.94) | 6.79 (1.12)
  Days 29 and 30 (n = 5, 5) | 6.44 (1.09) | 6.42 (0.79)
  Days 57 and 58 (n = 5, 5) | 6.36 (0.88) | 6.94 (0.94)
  Days 88 and 90 (n = 5, 5) | 5.98 (1.24) | 6.34 (0.75)
  1 wk postdose (n = 5, 5) | 6.1 (1.51) | 7.1 (1.78)
  2 wk postdose (n = 5, 5) | 6.34 (0.92) | 6.42 (0.46)

10. Secondary Outcome: Red Blood Cell (RBC) Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: Participants that completed three months of cobalt supplementation. Individual male baseline values for the 1-wk predose draw and the day 1 (predose) draw were averaged together. For females, the average baseline is the 1-wk predose data only because there was a significant difference between the 1-wk predose draw and the day 1 (predose) draw.
Measure: Mean (Standard Deviation); unit: million cells/µL
Groups:
- Female RBC: RBC levels before, during and after dosing
- Male RBC: RBC levels before, during, and after dosing
Arm/Group | Female RBC | Male RBC
Number analyzed (Participants) | 5 | 5
million cells/µL
  Baseline (n = 5, 5) | 4.42 (0.28) | 4.71 (0.2)
  Days 29 and 30 (n = 5, 5) | 4.28 (0.18) | 4.70 (0.20)
  Days 57 and 58 (n = 5, 5) | 4.3 (0.21) | 4.81 (0.18)
  Days 88 and 90 (n = 5, 5) | 4.32 (0.27) | 4.72 (0.32)
  1 wk postdose (n = 5, 5) | 4.42 (0.37) | 4.77 (0.24)
  2 wk postdose (n = 5, 5) | 4.38 (0.31) | 4.79 (0.21)

11. Secondary Outcome: Hematocrit Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Female Hematocrit: Hematocrit levels before, during and after dosing
- Male Hematocrit: Hematocrit levels before, during, and after dosing
Arm/Group | Female Hematocrit | Male Hematocrit
Number analyzed (Participants) | 5 | 5
Percentage
  Baseline (n = 5, 5) | 41.5 (1.68) | 45.1 (2.53)
  Days 29 and 30 (n = 5, 5) | 40.9 (1.15) | 45.0 (2.54)
  Days 57 and 58 (n = 5, 5) | 41.0 (1.14) | 46.3 (2.75)
  Days 88 and 90 (n = 5, 5) | 40.9 (2.00) | 45.0 (2.9)
  1 wk postdose (n = 5, 5) | 41.7 (2.17) | 45.8 (2.39)
  2 wk postdose (n = 5, 5) | 40.9 (2.42) | 45.7 (1.11)

12. Secondary Outcome: Protein Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Female Protein: Protein levels before, during and after dosing
- Male Protein: Protein levels before, during, and after dosing
Arm/Group | Female Protein | Male Protein
Number analyzed (Participants) | 5 | 5
g/dL
  Baseline (n = 5, 5) | 7.11 (0.33) | 7.26 (0.30)
  Days 29 and 30 (n = 5, 5) | 7.00 (0.35) | 7.24 (0.30)
  Days 57 and 58 (n = 5, 5) | 7.08 (0.28) | 7.16 (0.31)
  Days 88 and 90 (n = 5, 5) | 7.02 (0.38) | 7.14 (0.11)
  1 wk postdose (n = 5, 5) | 6.96 (0.48) | 7.28 (0.33)
  2 wk postdose (n =5, 5) | 7.04 (0.29) | 7.32 (0.41)

13. Secondary Outcome: Albumin Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Female Albumin: Albumin levels before, during and after dosing
- Male Albumin: Albumin levels before, during, and after dosing
Arm/Group | Female Albumin | Male Albumin
Number analyzed (Participants) | 5 | 5
g/dL
  Baseline (n = 5, 5) | 4.39 (0.22) | 4.63 (0.32)
  Days 29 and 30 (n = 5, 5) | 4.32 (0.16) | 4.60 (0.37)
  Days 57 and 58 (n = 5, 5) | 4.34 (0.17) | 4.56 (0.23)
  Days 88 and 90 (n = 5, 5) | 4.28 (0.19) | 4.48 (0.25)
  1 wk postdose (n = 5, 5) | 4.20 (0.27) | 4.60 (0.3)
  2 wk postdose (n = 5, 5) | 4.32 (0.25) | 4.56 (0.3)

14. Secondary Outcome: Thyroid-Stimulating Hormone (TSH) Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mIU/L
Groups:
- Female TSH: TSH levels before, during and after dosing
- Male TSH: TSH levels before, during, and after dosing
Arm/Group | Female TSH | Male TSH
Number analyzed (Participants) | 5 | 5
mIU/L
  Baseline (n = 5, 5) | 1.73 (0.77) | 2.35 (1.72)
  Days 29 and 30 (n = 5, 5) | 1.53 (1.03) | 3.35 (3.82)
  Days 57 and 58 (n = 5, 5) | 1.65 (1.08) | 3.11 (3.65)
  Days 88 and 90 (n = 5, 5) | 2.30 (1.90) | 2.24 (2.02)
  1 wk postdose (n = 5, 5) | 1.73 (0.90) | 2.30 (1.93)
  2 wk postdose (n = 5, 5) | 1.55 (0.63) | 2.33 (2.35)

15. Secondary Outcome: T4 Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: Participants that completed three months of cobalt supplementation.Individual baseline values for the 1-wk predose draw and the day 1 (predose) draw were averaged together to give one baseline value.
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Female T4: T4 levels before, during and after dosing
- Male T4: T4 levels before, during, and after dosing
Arm/Group | Female T4 | Male T4
Number analyzed (Participants) | 5 | 5
ng/dL
  Baseline (n = 5, 5) | 1.10 (0.11) | 1.15 (0.15)
  Days 29 and 30 (n = 5, 5) | 1.16 (0.11) | 1.16 (0.13)
  Days 57 and 58 (n = 5, 5) | 1.12 (0.11) | 1.16 (0.13)
  Days 88 and 90 (n = 5, 5) | 1.08 (0.18) | 1.12 (0.08)
  1 wk postdose (n = 5, 5) | 1.22 (0.13) | 1.15 (0.10)
  2 wk postdose (n = 5, 5) | 1.06 (0.11) | 1.14 (0.05)

16. Secondary Outcome: Total Iron Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg/dL
Groups:
- Female Total Iron: Total iron levels before, during and after dosing
- Male Total Iron: Total iron levels before, during, and after dosing
Arm/Group | Female Total Iron | Male Total Iron
Number analyzed (Participants) | 5 | 5
µg/dL
  Baseline (n = 5, 5) | 88.4 (12.6) | 122 (26.4)
  Days 29 and 30 (n = 5, 5) | 77.4 (21.5) | 119 (39.5)
  Days 57 and 58 (n = 5, 5) | 84.6 (19.4) | 105 (47.1)
  Days 88 and 90 (n = 5, 5) | 79.2 (21) | 82.6 (32.6)
  1 wk postdose (n = 5, 5) | 77.6 (51.4) | 115 (37.1)
  2 wk postdose (n = 5, 5) | 64 (11.6) | 111 (42.8)

17. Secondary Outcome: Ferritin Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: Participants that completed three months of cobalt supplementation. Individual female baseline values for the 1-wk predose draw and the day 1 (predose) draw were averaged together. For males, the average baseline is the 1-wk predose data only because there was a significant difference between the 1-wk predose draw and the day 1 (predose) draw.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Female Ferritin: Ferritin levels before, during and after dosing
- Male Ferritin: Ferritin levels before, during, and after dosing
Arm/Group | Female Ferritin | Male Ferritin
Number analyzed (Participants) | 5 | 5
ng/mL
  Baseline (n = 5, 5) | 51.3 (40.4) | 136 (77.3)
  Days 29 and 30 (n = 5, 5) | 32.0 (24.2) | 95.2 (57.5)
  Days 57 and 58 (n = 5, 5) | 27.4 (23.2) | 86.6 (59.6)
  Days 88 and 90 (n = 5, 5) | 21.6 (14.7) | 85.2 (53.1)
  1 wk postdose (n = 5, 5) | 34.6 (43.4) | 74.6 (50.3)
  2 wk postdose (n = 5, 5) | 24.8 (18.7) | 90.4 (66.0)

18. Secondary Outcome: Creatine Creatine Kinase-Myocardial Band (CK-MB) Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Female CK-MB: CK-MB levels before, during and after dosing
- Male CK-MB: CK-MB levels before, during, and after dosing
Arm/Group | Female CK-MB | Male CK-MB
Number analyzed (Participants) | 5 | 5
ng/mL
  Baseline (n = 5, 5) | 0.61 (0.37) | 1.58 (0.68)
  Days 29 and 30 (n = 5, 5) | 0.80 (0.45) | 0.97 (0.95)
  Days 57 and 58 (n = 5, 5) | 0.59 (0.35) | 0.92 (0.85)
  Days 88 and 90 (n = 5, 5) | 1.03 (0.56) | 1.23 (0.82)
  1 wk postdose (n = 5, 5) | 0.81 (0.36) | 1.25 (1.08)
  2 wk postdose (n = 5, 5) | 1.09 (0.48) | 1.42 (1.53)

19. Secondary Outcome: Creatinine Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Female Creatine: Creatine levels before, during and after dosing
- Male Creatine: Creatine levels before, during, and after dosing
Arm/Group | Female Creatine | Male Creatine
Number analyzed (Participants) | 5 | 5
mg/dL
  Baseline (n = 5, 5) | 0.79 (0.09) | 1.05 (0.09)
  Days 29 and 30 (n = 5, 5) | 0.78 (0.07) | 1.01 (0.16)
  Days 57 and 58 (n = 5, 5) | 0.77 (0.08) | 1.04 (0.11)
  Days 88 and 90 (n = 5, 5) | 0.80 (0.06) | 0.99 (0.10)
  1 wk postdose (n = 5, 5) | 0.84 (0.09) | 1.02 (0.12)
  2 wk postdose (n = 5, 5) | 0.82 (0.13) | 1.05 (0.10)

20. Secondary Outcome: Alanine Aminotransferase (ALT) Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Female ALT: ALT levels before, during and after dosing
- Male ALT: ALT levels before, during, and after dosing
Arm/Group | Female ALT | Male ALT
Number analyzed (Participants) | 5 | 5
U/L
  Baseline (n = 5, 5) | 14.8 (4.19) | 30.6 (19.3)
  Days 29 and 30 (n = 5, 5) | 13.6 (4.39) | 26.2 (13.5)
  Days 57 and 58 (n = 5, 5) | 14.8 (6.61) | 32.0 (19.3)
  Days 88 and 90 (n = 5, 5) | 11.2 (3.11) | 29.4 (17.1)
  1 wk postdose (n = 5, 5) | 12.6 (3.85) | 29.8 (15.6)
  2 wk postdose (n = 5, 5) | 15.8 (4.87) | 29.8 (14.5)

21. Secondary Outcome: Aspartate Aminotransferase (AST) Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Female AST: AST levels before, during and after dosing
- Male AST: AST levels before, during, and after dosing
Arm/Group | Female AST | Male AST
Number analyzed (Participants) | 5 | 5
U/L
  Baseline (n = 5, 5) | 18.8 (4.63) | 22.9 (4.26)
  Days 29 and 30 (n = 5, 5) | 17.6 (3.51) | 21.0 (4.06)
  Days 57 and 58 (n = 5, 5) | 20.2 (8.87) | 22.4 (7.02)
  Days 88 and 90 (n = 5, 5) | 15.8 (4.66) | 23.4 (6.5)
  1 wk postdose (n = 5, 5) | 16.8 (5.36) | 23.6 (4.72)
  2 wk postdose (n = 5, 5) | 20.6 (6.66) | 25.8 (9.60)

22. Secondary Outcome: HDL Cholesterol Levels After 3 Months of Cobalt Supplementation
Description: Blood chemistries assessed during the study included a lipid panel, comprehensive metabolic panel, creatine kinase-myocardial band, thyroid stimulating hormone, free thyroxine, and complete blood count with differential, total iron, and ferritin. HDL cholesterol levels were assessed before cobalt dietary supplementation and after three months of supplementation.
Time Frame: Study volunteers were assessed before and at the end of cobalt supplementation
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Female HDL Cholesterol; Male HDL Cholesterol: HDL cholesterol levels before and after cobalt supplementation
Arm/Group | Female HDL Cholesterol | Male HDL Cholesterol
Number analyzed (Participants) | 5 | 5
mg/dL
  Baseline | 85.2 (19.0) | 50.2 (14.1)
  Days 88 and 90 | 78.4 (23.1) | 50.6 (11.9)

23. Secondary Outcome: Total Cholesterol Levels After 3 Months of Cobalt Supplementation
Description: Blood chemistries assessed during the study included a lipid panel, comprehensive metabolic panel, creatine kinase-myocardial band, thyroid stimulating hormone, free thyroxine, and complete blood count with differential, total iron, and ferritin. Total cholesterol levels were assessed before cobalt dietary supplementation and after three months of supplementation.
Time Frame: Study volunteers were assessed before and at the end of cobalt supplementation
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Female Total Cholesterol; Male Total Cholesterol: Total cholesterol levels before and after cobalt supplementation
Arm/Group | Female Total Cholesterol | Male Total Cholesterol
Number analyzed (Participants) | 5 | 5
mg/dL
  Baseline | 209 (31.7) | 179 (26.6)
  Days 88 and 90 | 220 (54.6) | 188 (46.6)

24. Secondary Outcome: Triglyceride Levels After 3 Months of Cobalt Supplementation
Description: Blood chemistries assessed during the study included a lipid panel, comprehensive metabolic panel, creatine kinase-myocardial band, thyroid stimulating hormone, free thyroxine, and complete blood count with differential, total iron, and ferritin. Triglyceride levels were assessed before cobalt dietary supplementation and after three months of supplementation.
Time Frame: Study volunteers were assessed before and at the end of cobalt supplementation
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Female Triglycerides; Male Triglycerides: Triglyceride levels before and after cobalt supplementation
Arm/Group | Female Triglycerides | Male Triglycerides
Number analyzed (Participants) | 5 | 5
mg/dL
  Baseline | 105 (41.3) | 113 (51.1)
  Days 88 and 90 | 95.6 (29.6) | 122 (71.5)

25. Secondary Outcome: Glucose Levels After 1, 2 and 3 Months of Dosing
Description: as for outcome 3
Time Frame: Study volunteers were assessed before, during and after cobalt supplementation (2 wk post)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Female Glucose: Glucose levels before, during and after dosing
- Male Glucose: Glucose levels before, during, and after dosing
Arm/Group | Female Glucose | Male Glucose
Number analyzed (Participants) | 5 | 5
mg/dL
  Baseline (n = 5, 5) | 88.2 (7.53) | 89.9 (13)
  Days 29 and 30 (n = 5, 5) | 82.2 (10.1) | 83.4 (9.76)
  Days 57 and 58 (n = 5, 5) | 86.4 (9.4) | 81.2 (26.1)
  Days 88 and 90 (n = 5, 5) | 83.2 (9.91) | 87.4 (13.8)
  1 wk postdose (n = 5, 5) | 79.6 (14.5) | 90.6 (2.97)
  2 wk postdose (n = 5, 5) | 88.4 (15.1) | 79.4 (9.5)

26. Secondary Outcome: Cobalt Urine Concentrations
Description: A 24 hr urine collection for cobalt analysis was performed at Day 14/16, Day 43/44 and Day 88/90.
Time Frame: During cobalt supplementation
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: µg/L
Groups:
- Female Cobalt Urine Concentrations; Male Cobalt Urine Concentrations: Cobalt urine concentrations during daily oral intake of 1 mg Co.
Arm/Group | Female Cobalt Urine Concentrations | Male Cobalt Urine Concentrations
Number analyzed (Participants) | 5 | 5
µg/L
  Day 14/16 | 186 (170) | 119 (114)
  Day 43/44 | 226 (228) | 46 (35)
  Day 88/90 | 193 (179) | 70 (29)

27. Secondary Outcome: Cobalt Urine Concentrations After Cessation of Cobalt Supplementation
Description: A 24 hr urine collection for cobalt analysis was performed on three volunteers (two females and one male) at one, two, six and ten weeks post-dosing. The one male volunteer provided three consecutive 24-hr urine samples at the one and two week post-dosing time points; data for individual urine collections were averaged together to give an average one and two week post-dosing data concentration.
Time Frame: After cobalt supplementation
Population: Participants that completed three months of cobalt supplementation and volunteered to do additional urine collections after stopping cobalt supplementation. "n" represents the number of urine samples analyzd at each time point.
Measure: Mean (Standard Deviation); unit: µg/L
Groups:
- Female Cobalt Urine Concentrations; Male Cobalt Urine Concentrations: Cobalt urine concentrations after cessation of cobalt supplementation
Arm/Group | Female Cobalt Urine Concentrations | Male Cobalt Urine Concentrations
Number analyzed (Participants) | 2 | 1
µg/L
  1 wk postdose (n = 5, 3) | 38 (29) | 14 (6)
  2 wk postdose (n = 4, 3) | 19 (18) | 7 (2)
  6 wk postdose (n = 2, 1) | 6 (5) | 2 (0)
  10 wk postdose (n = 2, 1) | 6 (7) | 1 (0)

28. Primary Outcome: Cobalt Serum Concentrations
Description: as for outcome 8
Time Frame: Before, during and after cobalt supplementation
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: µg Co/L
Groups:
- Female Cobalt Serum Concentrations; Male Cobalt Serum Concentrations: Volunteers (males and females) were instructed to take the cobalt dietary supplement in the morning according to the manufacturer's label, which suggested a serving of 1 mg cobalt (~2 mL) daily "in water or juice as maintenance." Dietary supplementation lasted for approximately three months.
Arm/Group | Female Cobalt Serum Concentrations | Male Cobalt Serum Concentrations
Number analyzed (Participants) | 5 | 5
µg Co/L
  Day 4/5 | 23.3 (12.4) | 11.0 (5.7)
  Day 8/9 | 42.3 (33.4) | 11.8 (9.7)
  Day 14/16 | 42.5 (30.9) | 20.4 (11.5)
  Day 22/24 | 36.8 (24.2) | 34.7 (23.1)
  Day 29/30 | 53.9 (35.8) | 23.9 (8.7)
  Day 43/44 | 48.2 (34.5) | 24.3 (16.5)
  Day 57/58 | 34.9 (20.3) | 24.1 (15.7)
  Day 71/72 | 46.1 (40.8) | 28.2 (18.0)
  Day 88/90 | 71.2 (60.0) | 25.2 (13.2)
  1 wk post | 21.9 (20.6) | 8.4 (3.1)
  2 wk post | 12.5 (11.6) | 4.6 (1.6)
  6 wk post | 3.8 (3.3) | 1.4 (0.8)
  10 wk post | 1.9 (1.5) | 0.9 (0.4)
  4 month post | 0.96 (0.6) | 0.5 (0.3)

29. Secondary Outcome: Changes in Cardiac Function (LVEF)
Description: as for outcome 5
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: LVEF (2D est) (%)
Arm/Group | Prestudy | Study Midpoint | Study Completion
Number analyzed (Participants) | 10 | 10 | 10
LVEF (2D est) (%) | 65.9 (4.43) | 66.8 (4.21) | 65.0 (2.54)

30. Secondary Outcome: Changes in Cardiac Function (LA Volume Index)
Description: as for outcome 5
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: LA volume index (mL/m^2)
Arm/Group | Prestudy | Study Midpoint | Study Completion
Number analyzed (Participants) | 10 | 10 | 10
LA volume index (mL/m^2) | 23.3 (4.27) | 24.2 (5.33) | 24.0 (6.08)

31. Secondary Outcome: Changes in Visual Function (Average RNFL Thickness)
Description: as for outcome 6
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: Average RNFL thickness (µm)
Groups:
- Prestudy - Right; Study Midpoint - Right; Study Completion - Right: Values of the right eye for select RNFL variables
- Prestudy - Left; Study Midpoint - Left; Study Completion - Left: Values of the left eye for select RNFL variables
Arm/Group | Prestudy - Right | Prestudy - Left | Study Midpoint - Right | Study Midpoint - Left | Study Completion - Right | Study Completion - Left
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Average RNFL thickness (µm) | 97.10 (7.89) | 97.00 (8.67) | 97.00 (7.89) | 96.30 (8.64) | 96.50 (7.81) | 96.50 (9.01)

32. Secondary Outcome: Changes in Visual Function (Average C:D Ratio)
Description: as for outcome 6
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Prestudy - Right; Study Midpoint - Right; Study Completion - Right: Values of the right eye for select OHN variables
- Prestudy - Left; Study Midpoint - Left; Study Completion - Left: Values of the left eye for select OHN variables
Arm/Group | Prestudy - Right | Prestudy - Left | Study Midpoint - Right | Study Midpoint - Left | Study Completion - Right | Study Completion - Left
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ratio
  Average C:D ratio | 0.43 (0.12) | 0.44 (0.11) | 0.41 (0.13) | 0.42 (0.12) | 0.40 (0.12) | 0.40 (0.11)
  Vertical C:D ratio | 0.41 (0.13) | 0.40 (0.10) | 0.40 (0.12) | 0.39 (0.11) | 0.38 (0.13) | 0.36 (0.10)

33. Secondary Outcome: Changes in Visual Function (Cup Volume)
Description: as for outcome 6
Time Frame: Baseline, at the study midpoint, and at the study completion
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Prestudy - Right | Prestudy - Left | Study Midpoint - Right | Study Midpoint - Left | Study Completion - Right | Study Completion - Left
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
mm^3 | 0.09 (0.06) | 0.08 (0.04) | 0.08 (0.05) | 0.07 (0.04) | 0.08 (0.05) | 0.07 (0.04)

34. Secondary Outcome: Changes in Visual Function (VFI)
Description: as for outcome 6
Time Frame: Baseline, at the study midpoint, and at the study completion
Measure: Mean (Standard Deviation); unit: VFI (%)
Groups:
- Prestudy - Right; Study Midpoint - Right; Study Completion - Right: Values of the right eye for select VFI variables
- Prestudy - Left; Study Midpoint - Left; Study Completion - Left: Values of the left eye for select VFI variables
Arm/Group | Prestudy - Right | Prestudy - Left | Study Midpoint - Right | Study Midpoint - Left | Study Completion - Right | Study Completion - Left
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
VFI (%) | 99.40 (0.70) | 99.30 (0.82) | 99.30 (0.48) | 99.50 (0.97) | 99.60 (0.52) | 99.70 (0.48)

35. Secondary Outcome: Changes in Visual Function (Mean Deviation and PSD)
Description: as for outcome 6
Time Frame: Baseline, at the study midpoint, and at the study completion
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Prestudy - Right | Prestudy - Left | Study Midpoint - Right | Study Midpoint - Left | Study Completion - Right | Study Completion - Left
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
dB
  Mean deviation (dB) | -0.22 (1.01) | -0.25 (0.78) | 0.29 (0.85) | 0.02 (0.69) | 0.26 (0.82) | -0.09 (0.89)
  PSD (dB) | 1.44 (0.31) | 1.38 (0.30) | 1.37 (0.30) | 1.28 (0.13) | 1.26 (0.16) | 1.26 (0.16)

36. Secondary Outcome: Changes in Neurological Function (Sural Sensory Amplitude)
Description: as for outcome 7
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: Sural Sensory Amplitude (µV)
Groups:
- 1 mo Postdose: Values of the sural sensory and peroneal motor variables
Arm/Group | Prestudy | Study Midpoint | Study Completion | 1 mo Postdose
Number analyzed (Participants) | 10 | 10 | 10 | 10
Sural Sensory Amplitude (µV) | 24.2 (14.8) | 23.4 (14.9) | 20.7 (12.4) | 28.3 (24.2)

37. Secondary Outcome: Changes in Neurological Function (Velocity)
Description: as for outcome 7
Time Frame: Baseline, at the study midpoint, and at the study completion
Population: Participants that completed three months of cobalt supplementation
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Prestudy | Study Midpoint | Study Completion | 1 mo Postdose
Number analyzed (Participants) | 10 | 10 | 10 | 10
m/s
  Sural Sensory Velocity | 42.4 (5.8) | 39.9 (7.4) | 36.4 (7.0) | 43.3 (7.8)
  Peroneal Motor Velocity | 58.7 (13.7) | 64.1 (18.7) | 63.2 (24.8) | 0 (0)

ADVERSE EVENTS:
Time Frame: During the study: 7-8 months (approximate length of the study)
Description: Summary of self-reported adverse events
Groups:
- Study Volunteers: Study volunteers (males and females) were instructed to take the cobalt dietary supplement in the morning according to the manufacturer's label, which suggested a serving of 1 mg cobalt (~2 mL) daily "in water or juice as maintenance." Dietary supplementation lasted for approximately three months.
Arm/Group | Study Volunteers
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Volunteers (N=13)
Ear pain and tinnitus associated with sinusitis (General disorders) | 1 — The tinnitus persisted in the right ear throughout the remainder of the study and post-dosing period, but did not impact daily activities. At two months post-dosing, the volunteer still reported mild tinnitus on the side of his prior infection.
Migraine headaches with prior history of headache (General disorders) | 1 — The volunteer had a history of migraine headaches, and developed worsening headaches one week after starting to take the Co dietary supplement.
Vesicular rash following vaccination (General disorders) | 1 — The volunteer had recently received a tetanus vaccination, as well as other vaccinations for yellow fever and typhoid near the time of the rash development
Rash on face, neck, upper trunk, and back with peeling skin on palms of hands on both sides (General disorders) | 1 — Study leaders were notified approximately 72 hours after the rash first developed, and some of her symptoms had resolved by the time she was assessed by the study director. Her skin changes gradually resolved about a month after she stopped taking Co

LIMITATIONS AND CAVEATS:
The primary limitation of our study was its small sample size. We believe the study was sufficiently robust because we evaluated effects on hematologic and thyroid variables, both of which have been identified as sensitive markers of cobalt exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes